CLINICAL TRIAL: NCT01071382
Title: Epidemiology of Aeromedical Evacuation
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Workers Samaritan Federation Germany (Unknown)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: 002
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Apoplexy; Femoral Neck Fracture; Myocardial Infarction; Subarachnoid Hemorrhage; Polytrauma
Keywords: Aeromedical Evacuation; Repatriation
MeSH Terms: conditions — Stroke; Femoral Neck Fractures; Myocardial Infarction; Subarachnoid Hemorrhage; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Increasing air travel has resulted in a significant increase in aeromedical evacuation over the past decade. However there is only a small amount of epidemiological data available on the diagnosis, costs and transport characteristics of aeromedical evacuation cases. In the present study Cases of aeromedical evacuation by a relief organization (Workers' Samaritan Federation Germany) were analyzed based on the following criteria: age, sex and diagnosis of the patient, ventilation mode, days of illness before transport, type of transport, flight routes, flying time, flight distance, type of aircraft, type and distance of connecting transport from the destination airport to the final hospital, total cost per repatriation, and costs per flight-minute of each transport type.

ELIGIBILITY:
Inclusion Criteria:

* medical emergency and aeromedical evacuation / repatriation

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were repatriated from abroad because of a medical emergency
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Sand, Principal Investigator — Dermatologic Surgery Unit, Department of Dermatology and Allergology, Ruhr-University Bochum, Germany; PD Dr. Falk G. Bechara, Study Director — Dermatologic Surgery Unit, Department of Dermatology and Allergology, Ruhr-University Bochum, Germany; Univ.- Prof. Dr. Peter Altmeyer, Study Chair — Department of Dermatology and Allergology, Ruhr-University Bochum, Germany

REFERENCES:
- [Result] Sand M, Bollenbach M, Sand D, Lotz H, Thrandorf C, Cirkel C, Altmeyer P, Bechara FG. Epidemiology of aeromedical evacuation: an analysis of 504 cases. J Travel Med. 2010 Nov-Dec;17(6):405-9. doi: 10.1111/j.1708-8305.2010.00454.x. PMID 21050322